CLINICAL TRIAL: NCT00909038
Title: A Descriptive Pharmaco-epidemiological Study of a Hypertensive Patient Population Treated With a Fixed-dose Combination of Telmisartan 80 mg and Hydrochlorothiazide 25 mg and of Conditions for the Management of Arterial Hypertension
Brief Title: Telmisartan 80mg+Hydrochlorothiazide (HCTZ) 25 mg in Hypertension: an Observational Study
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.574
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2011-04-14 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
It is a national, retrospective , observational study in hypertensive patients treated for at least 8 weeks with the fixed dose combination of telmisartan 80 mg and hydrochlorothiazide 25 mg. The primary objective is to assess the control rate (systolic and diastolic blood pressure). Key secondary objectives are to assess the blood pressure reduction after at least 8 weeks of treatment, describe the population treated with this new fixed dose combination

ELIGIBILITY:
Inclusion criteria:

* Hypertensives
* Treated for at least 8 weeks with the fixed dose combination of telmisartan 80 mg and hydrochlorothiazide 25 mg

Exclusion criteria:

- Treated with the combination less than 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3440
Sampling Method: Probability Sample
Enrollment: 2411 (Actual)
Dates: Start 2009-05; Primary Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (915):
- France (915):
  - Boehringer Ingelheim Investigator site 1, Ablon-sur-Seine
  - Boehringer Ingelheim Investigator site 2, Achenheim
  - Boehringer Ingelheim Investigator site 3, Afa
  - Boehringer Ingelheim Investigator site 4, Aiguillon
  - Boehringer Ingelheim Investigator site 5, Aire-sur-l'Adour
  - Boehringer Ingelheim Investigator site 6, Aix-en-Othe
  - Boehringer Ingelheim Investigator site 7, Aix-en-Provence
  - Boehringer Ingelheim Investigator site 8, Aix-en-Provence
  - Boehringer Ingelheim Investigator site 9, Aix-les-Bains
  - Boehringer Ingelheim Investigator site 10, Ajaccio
  - Boehringer Ingelheim Investigator site 11, Ajaccio
  - Boehringer Ingelheim Investigator site 12, Amagne
  - Boehringer Ingelheim Investigator site 13, Amiens
  - Boehringer Ingelheim Investigator site 14, Amiens
  - Boehringer Ingelheim Investigator site 15, Andard
  - Boehringer Ingelheim Investigator site 16, Angers
  - Boehringer Ingelheim Investigator site 17, Angoulême
  - Boehringer Ingelheim Investigator site 18, Angoulême
  - Boehringer Ingelheim Investigator site 19, Angoulême
  - Boehringer Ingelheim Investigator site 20, Annecy
  - Boehringer Ingelheim Investigator site 21, Annecy
  - Boehringer Ingelheim Investigator site 22, Annemasse
  - Boehringer Ingelheim Investigator site 23, Annonay
  - Boehringer Ingelheim Investigator site 24, Annonay
  - Boehringer Ingelheim Investigator site 25, Antibes
  - Boehringer Ingelheim Investigator site 26, Antony
  - Boehringer Ingelheim Investigator site 27, Anvin
  - Boehringer Ingelheim Investigator site 28, Anzin
  - Boehringer Ingelheim Investigator site 29, Appoigny
  - Boehringer Ingelheim Investigator site 30, Ardentes
  - Boehringer Ingelheim Investigator site 31, Argenteuil
  - Boehringer Ingelheim Investigator site 32, Arles
  - Boehringer Ingelheim Investigator site 33, Arques-la-Bataille
  - Boehringer Ingelheim Investigator site 34, Arradon
  - Boehringer Ingelheim Investigator site 35, Ars
  - Boehringer Ingelheim Investigator site 36, Arsac
  - Boehringer Ingelheim Investigator site 37, Artigues-près-Bordeaux
  - Boehringer Ingelheim Investigator site 38, Asnières-sur-Seine
  - Boehringer Ingelheim Investigator site 39, Asson
  - Boehringer Ingelheim Investigator site 40, Aubervilliers
  - Boehringer Ingelheim Investigator site 41, Auch
  - Boehringer Ingelheim Investigator site 42, Augny
  - Boehringer Ingelheim Investigator site 43, Aulnay-sous-Bois
  - Boehringer Ingelheim Investigator site 44, Aulnay-sous-Bois
  - Boehringer Ingelheim Investigator site 45, Aumetz
  - Boehringer Ingelheim Investigator site 46, Auxerre
  - Boehringer Ingelheim Investigator site 47, Auzon
  - Boehringer Ingelheim Investigator site 48, Avallon
  - Boehringer Ingelheim Investigator site 49, Bagneux
  - Boehringer Ingelheim Investigator site 50, Bagnols-sur-Cèze
  - Boehringer Ingelheim Investigator site 51, Baillet-en-France
  - Boehringer Ingelheim Investigator site 52, Bailleul
  - Boehringer Ingelheim Investigator site 53, Barbezieux-Saint-Hilaire
  - Boehringer Ingelheim Investigator site 54, Barbezieux-Saint-Hilaire
  - Boehringer Ingelheim Investigator site 55, Bassillac
  - Boehringer Ingelheim Investigator site 56, Bassussarry
  - Boehringer Ingelheim Investigator site 57, Bauvin
  - Boehringer Ingelheim Investigator site 58, Bayeux
  - Boehringer Ingelheim Investigator site 59, Beaumont-sur-Lèze
  - Boehringer Ingelheim Investigator site 60, Beauvais
  - Boehringer Ingelheim Investigator site 62, Belley
  - Boehringer Ingelheim Investigator site 63, Benfeld
  - Boehringer Ingelheim Investigator site 64, Bergerac
  - Boehringer Ingelheim Investigator site 65, Bergues
  - Boehringer Ingelheim Investigator site 66, Bersée
  - Boehringer Ingelheim Investigator site 61, Bélâbre
  - Boehringer Ingelheim Investigator site 67, Béthisy-Saint-Pierre
  - Boehringer Ingelheim Investigator site 68, Béziers
  - Boehringer Ingelheim Investigator site 69, Biarritz
  - Boehringer Ingelheim Investigator site 70, Biganos
  - Boehringer Ingelheim Investigator site 71, Biganos
  - Boehringer Ingelheim Investigator site 72, Biganos
  - Boehringer Ingelheim Investigator site 73, Billère
  - Boehringer Ingelheim Investigator site 74, Billère
  - Boehringer Ingelheim Investigator site 75, Blangy-sur-Bresle
  - Boehringer Ingelheim Investigator site 76, Blanquefort
  - Boehringer Ingelheim Investigator site 77, Blaye
  - Boehringer Ingelheim Investigator site 78, Bleriot
  - Boehringer Ingelheim Investigator site 79, Blois
  - Boehringer Ingelheim Investigator site 80, Blotzheim
  - Boehringer Ingelheim Investigator site 81, Bohain-en-Vermandois
  - Boehringer Ingelheim Investigator site 82, Bois-Colombes
  - Boehringer Ingelheim Investigator site 83, Bois-Colombes
  - Boehringer Ingelheim Investigator site 84, Boiscommun
  - Boehringer Ingelheim Investigator site 85, Bondoufle
  - Boehringer Ingelheim Investigator site 86, Bondoufle
  - Boehringer Ingelheim Investigator site 87, Bondues
  - Boehringer Ingelheim Investigator site 88, Boos
  - Boehringer Ingelheim Investigator site 89, Boos
  - Boehringer Ingelheim Investigator site 90, Bordeaux
  - Boehringer Ingelheim Investigator site 91, Bordeaux
  - Boehringer Ingelheim Investigator site 92, Bordeaux
  - Boehringer Ingelheim Investigator site 93, Bordeaux
  - Boehringer Ingelheim Investigator site 94, Bouilly
  - Boehringer Ingelheim Investigator site 95, Boulogne-Billancourt
  - Boehringer Ingelheim Investigator site 96, Bourg-la-Reine
  - Boehringer Ingelheim Investigator site 97, Bourron-Marlotte
  - Boehringer Ingelheim Investigator site 98, Bourth
  - Boehringer Ingelheim Investigator site 99, Braine
  - Boehringer Ingelheim Investigator site 100, Brest
  - Boehringer Ingelheim Investigator site 101, Brest
  - Boehringer Ingelheim Investigator site 102, Brest
  - Boehringer Ingelheim Investigator site 103, Brest
  - Boehringer Ingelheim Investigator site 104, Brest
  - Boehringer Ingelheim Investigator site 105, Bretenoux
  - Boehringer Ingelheim Investigator site 107, Breteuil
  - Boehringer Ingelheim Investigator site 106, Breteuil
  - Boehringer Ingelheim Investigator site 108, Bretignolles-sur-Mer
  - Boehringer Ingelheim Investigator site 109, Bretteville-l'Orgueilleuse
  - Boehringer Ingelheim Investigator site 110, Brie
  - Boehringer Ingelheim Investigator site 111, Brienne-le-Château
  - Boehringer Ingelheim Investigator site 112, Briouze
  - Boehringer Ingelheim Investigator site 113, Bron
  - Boehringer Ingelheim Investigator site 114, Bruère-Allichamps
  - Boehringer Ingelheim Investigator site 115, Bruges
  - Boehringer Ingelheim Investigator site 116, Brunehamel
  - Boehringer Ingelheim Investigator site 117, Buchy
  - Boehringer Ingelheim Investigator site 118, Bulgnéville
  - Boehringer Ingelheim Investigator site 119, Bulgnéville
  - Boehringer Ingelheim Investigator site 120, Cabanac-et-Villagrains
  - Boehringer Ingelheim Investigator site 121, Cabannes
  - Boehringer Ingelheim Investigator site 122, Cabestany
  - Boehringer Ingelheim Investigator site 123, Caen
  - Boehringer Ingelheim Investigator site 124, Cagnes-sur-Mer
  - Boehringer Ingelheim Investigator site 125, Cagnes-sur-Mer
  - Boehringer Ingelheim Investigator site 126, Cagnes-sur-Mer
  - Boehringer Ingelheim Investigator site 127, Callac de Bretagne
  - Boehringer Ingelheim Investigator site 128, Callac de Bretagne
  - Boehringer Ingelheim Investigator site 129, Cancon
  - Boehringer Ingelheim Investigator site 130, Canéjan
  - Boehringer Ingelheim Investigator site 131, Cannes
  - Boehringer Ingelheim Investigator site 132, Cannes
  - Boehringer Ingelheim Investigator site 133, Cannes
  - Boehringer Ingelheim Investigator site 134, Cany-Barville
  - Boehringer Ingelheim Investigator site 135, Capdenac-Gare
  - Boehringer Ingelheim Investigator site 136, Capdenac-Gare
  - Boehringer Ingelheim Investigator site 137, Carbon-Blanc
  - Boehringer Ingelheim Investigator site 138, Carcassonne
  - Boehringer Ingelheim Investigator site 139, Carcassonne
  - Boehringer Ingelheim Investigator site 140, Carcassonne
  - Boehringer Ingelheim Investigator site 141, Carhaix-Plouguer
  - Boehringer Ingelheim Investigator site 142, Carpentras
  - Boehringer Ingelheim Investigator site 143, Carvin
  - Boehringer Ingelheim Investigator site 144, Cassis
  - Boehringer Ingelheim Investigator site 145, Castanet-Tolosan
  - Boehringer Ingelheim Investigator site 146, Castelnau-le-Lez
  - Boehringer Ingelheim Investigator site 147, Castelsarrasin
  - Boehringer Ingelheim Investigator site 148, Castelsarrasin
  - Boehringer Ingelheim Investigator site 149, Castets
  - Boehringer Ingelheim Investigator site 150, Castets-en-Dorthe
  - Boehringer Ingelheim Investigator site 151, Cavalaire-sur-Mer
  - Boehringer Ingelheim Investigator site 152, Cepoy
  - Boehringer Ingelheim Investigator site 153, Cergy
  - Boehringer Ingelheim Investigator site 155, Cernay
  - Boehringer Ingelheim Investigator site 154, Cérilly
  - Boehringer Ingelheim Investigator site 157, Chalais
  - Boehringer Ingelheim Investigator site 158, Chambray-lès-Tours
  - Boehringer Ingelheim Investigator site 159, Champs-sur-Marne
  - Boehringer Ingelheim Investigator site 160, Chantilly
  - Boehringer Ingelheim Investigator site 161, Chaource
  - Boehringer Ingelheim Investigator site 162, Charleville-Mézières
  - Boehringer Ingelheim Investigator site 163, Charleville-Mézières
  - Boehringer Ingelheim Investigator site 164, Chassieu
  - Boehringer Ingelheim Investigator site 171, Chateauneuf Ille Vilaine
  - Boehringer Ingelheim Investigator site 176, Chaumont
  - Boehringer Ingelheim Investigator site 177, Chauvigny
  - Boehringer Ingelheim Investigator site 178, Chauvigny
  - Boehringer Ingelheim Investigator site 179, Chauvigny
  - Boehringer Ingelheim Investigator site 156, Châbons
  - Boehringer Ingelheim Investigator site 165, Château-Chinon(Ville)
  - Boehringer Ingelheim Investigator site 166, Château-d'Olonne
  - Boehringer Ingelheim Investigator site 167, Château-Renault
  - Boehringer Ingelheim Investigator site 168, Château-Thébaud
  - Boehringer Ingelheim Investigator site 169, Châteaubernard
  - Boehringer Ingelheim Investigator site 170, Châteaubriant
  - Boehringer Ingelheim Investigator site 172, Châteauroux
  - Boehringer Ingelheim Investigator site 173, Châtenay-Malabry
  - Boehringer Ingelheim Investigator site 174, Châtillon-Coligny
  - Boehringer Ingelheim Investigator site 175, Châtillon-sur-Seine
  - Boehringer Ingelheim Investigator site 180, Chelles
  - Boehringer Ingelheim Investigator site 181, Cherves-Richemont
  - Boehringer Ingelheim Investigator site 182, Chinon
  - Boehringer Ingelheim Investigator site 183, Claira
  - Boehringer Ingelheim Investigator site 184, Clamart
  - Boehringer Ingelheim Investigator site 185, Claye-Souilly
  - Boehringer Ingelheim Investigator site 186, Clermont-Ferrand
  - Boehringer Ingelheim Investigator site 187, Clichy
  - Boehringer Ingelheim Investigator site 188, Clisson
  - Boehringer Ingelheim Investigator site 189, Cognac
  - Boehringer Ingelheim Investigator site 190, Colombes
  - Boehringer Ingelheim Investigator site 191, Colombes
  - Boehringer Ingelheim Investigator site 192, Colombes
  - Boehringer Ingelheim Investigator site 193, Combles
  - Boehringer Ingelheim Investigator site 194, Comines
  - Boehringer Ingelheim Investigator site 195, Condé-sur-l'Escaut
  - Boehringer Ingelheim Investigator site 196, Condom
  - Boehringer Ingelheim Investigator site 197, Conflans Ste Honorine
  - Boehringer Ingelheim Investigator site 198, Conflans Ste Honorine
  - Boehringer Ingelheim Investigator site 199, Corbehem
  - Boehringer Ingelheim Investigator site 200, Cornebarrieu
  - Boehringer Ingelheim Investigator site 201, Coubron
  - Boehringer Ingelheim Investigator site 202, Courbevoie
  - Boehringer Ingelheim Investigator site 203, Courbevoie
  - Boehringer Ingelheim Investigator site 204, Courseulles-sur-Mer
  - Boehringer Ingelheim Investigator site 205, Coutances
  - Boehringer Ingelheim Investigator site 206, Creil
  - Boehringer Ingelheim Investigator site 207, Creully
  - Boehringer Ingelheim Investigator site 208, Creutzwald
  - Boehringer Ingelheim Investigator site 209, Croix
  - Boehringer Ingelheim Investigator site 210, Croix
  - Boehringer Ingelheim Investigator site 211, Cros-de-Cagnes
  - Boehringer Ingelheim Investigator site 212, Crosne
  - Boehringer Ingelheim Investigator site 213, Cugnaux
  - Boehringer Ingelheim Investigator site 214, Culoz
  - Boehringer Ingelheim Investigator site 215, Damprichard
  - Boehringer Ingelheim Investigator site 216, Damvillers
  - Boehringer Ingelheim Investigator site 217, Danjoutin
  - Boehringer Ingelheim Investigator site 218, Dax
  - Boehringer Ingelheim Investigator site 219, Décines-Charpieu
  - Boehringer Ingelheim Investigator site 220, Diemeringen
  - Boehringer Ingelheim Investigator site 221, Digne-les-Bains
  - Boehringer Ingelheim Investigator site 222, Dijon
  - Boehringer Ingelheim Investigator site 223, Dijon
  - Boehringer Ingelheim Investigator site 224, Dijon
  - Boehringer Ingelheim Investigator site 225, Dinan
  - Boehringer Ingelheim Investigator site 226, Dinard
  - Boehringer Ingelheim Investigator site 227, Dole
  - Boehringer Ingelheim Investigator site 228, Domont
  - Boehringer Ingelheim Investigator site 229, Douai
  - Boehringer Ingelheim Investigator site 230, Dourdan
  - Boehringer Ingelheim Investigator site 231, Douvaine
  - Boehringer Ingelheim Investigator site 232, Douvres-la-Délivrande
  - Boehringer Ingelheim Investigator site 233, Drancy
  - Boehringer Ingelheim Investigator site 234, Drancy
  - Boehringer Ingelheim Investigator site 235, Drap
  - Boehringer Ingelheim Investigator site 236, Drulingen
  - Boehringer Ingelheim Investigator site 239, Elliant
  - Boehringer Ingelheim Investigator site 240, Enghien-les-Bains
  - Boehringer Ingelheim Investigator site 241, Enghien-les-Bains
  - Boehringer Ingelheim Investigator site 247, Ermont
  - Boehringer Ingelheim Investigator site 248, Esquerdes
  - Boehringer Ingelheim Investigator site 249, Estrablin
  - Boehringer Ingelheim Investigator site 250, Estrées-Saint-Denis
  - Boehringer Ingelheim Investigator site 252, Eu
  - Boehringer Ingelheim Investigator site 253, Eygalières
  - Boehringer Ingelheim Investigator site 254, Eyragues
  - Boehringer Ingelheim Investigator site 237, Échirolles
  - Boehringer Ingelheim Investigator site 238, Échirolles
  - Boehringer Ingelheim Investigator site 242, Épernay
  - Boehringer Ingelheim Investigator site 243, Épernon
  - Boehringer Ingelheim Investigator site 244, Épierre
  - Boehringer Ingelheim Investigator site 245, Épinal
  - Boehringer Ingelheim Investigator site 246, Épinay-sur-Orge
  - Boehringer Ingelheim Investigator site 251, Étampes
  - Boehringer Ingelheim Investigator site 255, Fabrezan
  - Boehringer Ingelheim Investigator site 256, Faches-Thumesnil
  - Boehringer Ingelheim Investigator site 257, Famars
  - Boehringer Ingelheim Investigator site 258, Fauquembergues
  - Boehringer Ingelheim Investigator site 259, Fécamp
  - Boehringer Ingelheim Investigator site 260, Félines
  - Boehringer Ingelheim Investigator site 261, Figeac
  - Boehringer Ingelheim Investigator site 262, Firmi
  - Boehringer Ingelheim Investigator site 263, Firminy
  - Boehringer Ingelheim Investigator site 264, Fitilieu
  - Boehringer Ingelheim Investigator site 265, Flayosc
  - Boehringer Ingelheim Investigator site 266, Fleurance
  - Boehringer Ingelheim Investigator site 267, Fleury-sur-Orne
  - Boehringer Ingelheim Investigator site 268, Flize
  - Boehringer Ingelheim Investigator site 269, Florensac
  - Boehringer Ingelheim Investigator site 270, Folembray
  - Boehringer Ingelheim Investigator site 271, Fontaine-lès-Dijon
  - Boehringer Ingelheim Investigator site 272, Fontaine-lès-Dijon
  - Boehringer Ingelheim Investigator site 273, Fontenay-le-Comte
  - Boehringer Ingelheim Investigator site 274, Fontenay-sous-Bois
  - Boehringer Ingelheim Investigator site 275, Fos-sur-Mer
  - Boehringer Ingelheim Investigator site 276, Fosses
  - Boehringer Ingelheim Investigator site 277, Fougères
  - Boehringer Ingelheim Investigator site 278, Fougères
  - Boehringer Ingelheim Investigator site 279, Franconville
  - Boehringer Ingelheim Investigator site 280, Frasne
  - Boehringer Ingelheim Investigator site 281, Frencq
  - Boehringer Ingelheim Investigator site 282, Fresnes-sur-Escaut
  - Boehringer Ingelheim Investigator site 283, Froideconche
  - Boehringer Ingelheim Investigator site 284, Fruges
  - Boehringer Ingelheim Investigator site 285, Gagny
  - Boehringer Ingelheim Investigator site 286, Gallardon
  - Boehringer Ingelheim Investigator site 287, Garchizy
  - Boehringer Ingelheim Investigator site 288, Gâvres
  - Boehringer Ingelheim Investigator site 289, Gennes
  - Boehringer Ingelheim Investigator site 290, Gentilly
  - Boehringer Ingelheim Investigator site 291, Giraumont
  - Boehringer Ingelheim Investigator site 292, Gironcourt-sur-Vraine
  - Boehringer Ingelheim Investigator site 293, Golbey
  - Boehringer Ingelheim Investigator site 294, Gondrecourt-le-Château
  - Boehringer Ingelheim Investigator site 295, Gontaud-de-Nogaret
  - Boehringer Ingelheim Investigator site 296, Goudelin
  - Boehringer Ingelheim Investigator site 297, Gouville-sur-Mer
  - Boehringer Ingelheim Investigator site 298, Grambois
  - Boehringer Ingelheim Investigator site 299, Gray
  - Boehringer Ingelheim Investigator site 300, Grenoble
  - Boehringer Ingelheim Investigator site 301, Grenoble
  - Boehringer Ingelheim Investigator site 302, Grenoble
  - Boehringer Ingelheim Investigator site 303, Grenoble
  - Boehringer Ingelheim Investigator site 304, Grenoble
  - Boehringer Ingelheim Investigator site 305, Grenoble
  - Boehringer Ingelheim Investigator site 306, Grignols
  - Boehringer Ingelheim Investigator site 307, Guémar
  - Boehringer Ingelheim Investigator site 308, Guignicourt
  - Boehringer Ingelheim Investigator site 309, Guilvinec
  - Boehringer Ingelheim Investigator site 310, Haguenau
  - Boehringer Ingelheim Investigator site 311, Ham
  - Boehringer Ingelheim Investigator site 312, Hanvec
  - Boehringer Ingelheim Investigator site 313, Harfleur
  - Boehringer Ingelheim Investigator site 314, Harnes
  - Boehringer Ingelheim Investigator site 315, Hayange
  - Boehringer Ingelheim Investigator site 316, Hégenheim
  - Boehringer Ingelheim Investigator site 317, Hossegor
  - Boehringer Ingelheim Investigator site 318, Houdan
  - Boehringer Ingelheim Investigator site 319, Hyères
  - Boehringer Ingelheim Investigator site 320, Igé
  - Boehringer Ingelheim Investigator site 321, Imphy
  - Boehringer Ingelheim Investigator site 322, Inchy
  - Boehringer Ingelheim Investigator site 323, Issoudun
  - Boehringer Ingelheim Investigator site 324, Issy-les-Moulineaux
  - Boehringer Ingelheim Investigator site 325, Istres
  - Boehringer Ingelheim Investigator site 326, Istres
  - Boehringer Ingelheim Investigator site 327, Istres
  - Boehringer Ingelheim Investigator site 328, Ivry-sur-Seine
  - Boehringer Ingelheim Investigator site 329, Jargeau
  - Boehringer Ingelheim Investigator site 330, Jarny
  - Boehringer Ingelheim Investigator site 331, Jarville-la-Malgrange
  - Boehringer Ingelheim Investigator site 332, Jenlain
  - Boehringer Ingelheim Investigator site 333, Jeumont
  - Boehringer Ingelheim Investigator site 334, Juan-les-Pins
  - Boehringer Ingelheim Investigator site 335, Jussey
  - Boehringer Ingelheim Investigator site 336, Kunheim
  - Boehringer Ingelheim Investigator site 337, L'Aigle
  - Boehringer Ingelheim Investigator site 339, L'Escarène
  - Boehringer Ingelheim Investigator site 340, L'Escarène
  - Boehringer Ingelheim Investigator site 341, L'Île-Rousse
  - Boehringer Ingelheim Investigator site 342, L'Île-Rousse
  - Boehringer Ingelheim Investigator site 343, La Celle-Saint-Cloud
  - Boehringer Ingelheim Investigator site 344, La Ferté-Milon
  - Boehringer Ingelheim Investigator site 345, La Ferté-Saint-Aubin
  - Boehringer Ingelheim Investigator site 346, La Flèche
  - Boehringer Ingelheim Investigator site 347, La Francheville
  - Boehringer Ingelheim Investigator site 348, La Garenne-Colombes
  - Boehringer Ingelheim Investigator site 349, La Grande-Motte
  - Boehringer Ingelheim Investigator site 350, La Grande-Motte
  - Boehringer Ingelheim Investigator site 351, La Mothe-Saint-Héray
  - Boehringer Ingelheim Investigator site 352, La Primaube
  - Boehringer Ingelheim Investigator site 353, La Ricamarie
  - Boehringer Ingelheim Investigator site 354, La Riche
  - Boehringer Ingelheim Investigator site 355, La Roche-sur-Yon
  - Boehringer Ingelheim Investigator site 356, La Rochelle
  - Boehringer Ingelheim Investigator site 357, La Sauve
  - Boehringer Ingelheim Investigator site 358, La Talaudière
  - Boehringer Ingelheim Investigator site 359, La Tour-du-Crieu
  - Boehringer Ingelheim Investigator site 360, La Turballe
  - Boehringer Ingelheim Investigator site 361, La Varenne-Saint-Hilaire
  - Boehringer Ingelheim Investigator site 362, La Varenne-Saint-Hilaire
  - Boehringer Ingelheim Investigator site 363, Labastide-Murat
  - Boehringer Ingelheim Investigator site 364, Lagnieu
  - Boehringer Ingelheim Investigator site 365, Lagord
  - Boehringer Ingelheim Investigator site 366, Lamalou-les-Bains
  - Boehringer Ingelheim Investigator site 367, Lamalou-les-Bains
  - Boehringer Ingelheim Investigator site 368, Lambersart
  - Boehringer Ingelheim Investigator site 369, Lambersart
  - Boehringer Ingelheim Investigator site 370, Lambersart
  - Boehringer Ingelheim Investigator site 371, Lambersart
  - Boehringer Ingelheim Investigator site 372, Lancieux
  - Boehringer Ingelheim Investigator site 373, Lanester
  - Boehringer Ingelheim Investigator site 374, Lanester
  - Boehringer Ingelheim Investigator site 375, Lannion
  - Boehringer Ingelheim Investigator site 376, Lanouaille
  - Boehringer Ingelheim Investigator site 377, Lanvollon
  - Boehringer Ingelheim Investigator site 338, LArbresle
  - Boehringer Ingelheim Investigator site 378, Larche
  - Boehringer Ingelheim Investigator site 379, Lathus-Saint-Rémy
  - Boehringer Ingelheim Investigator site 380, Launaguet
  - Boehringer Ingelheim Investigator site 381, Lavaur
  - Boehringer Ingelheim Investigator site 382, Lavelanet
  - Boehringer Ingelheim Investigator site 383, Le Barcarès
  - Boehringer Ingelheim Investigator site 384, Le Blanc-Mesnil
  - Boehringer Ingelheim Investigator site 385, Le Bois-dOingt
  - Boehringer Ingelheim Investigator site 386, Le Brusc
  - Boehringer Ingelheim Investigator site 387, Le Cannet
  - Boehringer Ingelheim Investigator site 388, Le Cannet
  - Boehringer Ingelheim Investigator site 389, Le Cannet
  - Boehringer Ingelheim Investigator site 390, Le Clion-sur-Mer
  - Boehringer Ingelheim Investigator site 391, Le Golfe Juan
  - Boehringer Ingelheim Investigator site 392, Le Grand-Lemps
  - Boehringer Ingelheim Investigator site 393, Le Grand-Quevilly
  - Boehringer Ingelheim Investigator site 394, Le Havre
  - Boehringer Ingelheim Investigator site 395, Le Lavandou
  - Boehringer Ingelheim Investigator site 396, Le Lude
  - Boehringer Ingelheim Investigator site 397, Le Mans
  - Boehringer Ingelheim Investigator site 398, Le Mans
  - Boehringer Ingelheim Investigator site 399, Le Mans
  - Boehringer Ingelheim Investigator site 400, Le Mans
  - Boehringer Ingelheim Investigator site 401, Le Perray-en-Yvelines
  - Boehringer Ingelheim Investigator site 402, Le Perray-en-Yvelines
  - Boehringer Ingelheim Investigator site 403, Le Petit-Quevilly
  - Boehringer Ingelheim Investigator site 404, Le Plessis-Bouchard
  - Boehringer Ingelheim Investigator site 405, Le Pontet
  - Boehringer Ingelheim Investigator site 406, Le Pradet
  - Boehringer Ingelheim Investigator site 407, Le Soler
  - Boehringer Ingelheim Investigator site 408, Le Temple-de-Bretagne
  - Boehringer Ingelheim Investigator site 409, Le Touvet
  - Boehringer Ingelheim Investigator site 412, Lembach
  - Boehringer Ingelheim Investigator site 414, Les Andelys
  - Boehringer Ingelheim Investigator site 415, Les Bordes-sur-Arize
  - Boehringer Ingelheim Investigator site 416, Les Clayes-sous-Bois
  - Boehringer Ingelheim Investigator site 417, Les Mureaux
  - Boehringer Ingelheim Investigator site 418, Les Sables-d'Olonne
  - Boehringer Ingelheim Investigator site 419, Les Sorinières
  - Boehringer Ingelheim Investigator site 420, Levallois-Perret
  - Boehringer Ingelheim Investigator site 421, Lezoux
  - Boehringer Ingelheim Investigator site 411, Lège-Cap-Ferret
  - Boehringer Ingelheim Investigator site 410, Lédignan
  - Boehringer Ingelheim Investigator site 413, Léon
  - Boehringer Ingelheim Investigator site 422, Liévin
  - Boehringer Ingelheim Investigator site 423, Liffré
  - Boehringer Ingelheim Investigator site 424, Lille
  - Boehringer Ingelheim Investigator site 425, Lille
  - Boehringer Ingelheim Investigator site 426, Lille
  - Boehringer Ingelheim Investigator site 427, Limoges
  - Boehringer Ingelheim Investigator site 428, Limoges
  - Boehringer Ingelheim Investigator site 429, Limoges
  - Boehringer Ingelheim Investigator site 430, Limoges
  - Boehringer Ingelheim Investigator site 431, Limoux
  - Boehringer Ingelheim Investigator site 432, Linxe
  - Boehringer Ingelheim Investigator site 434, Lognes
  - Boehringer Ingelheim Investigator site 435, Lognes
  - Boehringer Ingelheim Investigator site 436, Longages
  - Boehringer Ingelheim Investigator site 437, Longjumeau
  - Boehringer Ingelheim Investigator site 440, Longueau
  - Boehringer Ingelheim Investigator site 441, Longuenesse
  - Boehringer Ingelheim Investigator site 438, Longué-Jumelles
  - Boehringer Ingelheim Investigator site 439, Longué-Jumelles
  - Boehringer Ingelheim Investigator site 442, Lorient
  - Boehringer Ingelheim Investigator site 443, Lorient
  - Boehringer Ingelheim Investigator site 444, Loudes
  - Boehringer Ingelheim Investigator site 445, Lyon
  - Boehringer Ingelheim Investigator site 446, Lyon
  - Boehringer Ingelheim Investigator site 447, Lyon
  - Boehringer Ingelheim Investigator site 448, Lyon
  - Boehringer Ingelheim Investigator site 433, Lœuilly
  - Boehringer Ingelheim Investigator site 449, Mably
  - Boehringer Ingelheim Investigator site 450, Magnac-Bourg
  - Boehringer Ingelheim Investigator site 451, Maisons-Alfort
  - Boehringer Ingelheim Investigator site 452, Maisons-Alfort
  - Boehringer Ingelheim Investigator site 453, Malicorne-sur-Sarthe
  - Boehringer Ingelheim Investigator site 454, Mantes-la-Ville
  - Boehringer Ingelheim Investigator site 455, Marcq-en-Barœul
  - Boehringer Ingelheim Investigator site 456, Mareuil-sur-Lay-Dissais
  - Boehringer Ingelheim Investigator site 457, Marignane
  - Boehringer Ingelheim Investigator site 458, Marlenheim
  - Boehringer Ingelheim Investigator site 459, Marmande
  - Boehringer Ingelheim Investigator site 460, Marquillies
  - Boehringer Ingelheim Investigator site 461, Marquillies
  - Boehringer Ingelheim Investigator site 462, Marseille
  - Boehringer Ingelheim Investigator site 463, Marseille
  - Boehringer Ingelheim Investigator site 464, Marseille
  - Boehringer Ingelheim Investigator site 465, Marseille
  - Boehringer Ingelheim Investigator site 466, Marseille
  - Boehringer Ingelheim Investigator site 467, Marseille
  - Boehringer Ingelheim Investigator site 468, Marseille
  - Boehringer Ingelheim Investigator site 469, Marseille
  - Boehringer Ingelheim Investigator site 470, Marseille
  - Boehringer Ingelheim Investigator site 471, Marseille
  - Boehringer Ingelheim Investigator site 472, Marseille
  - Boehringer Ingelheim Investigator site 473, Marseille
  - Boehringer Ingelheim Investigator site 474, Marseille
  - Boehringer Ingelheim Investigator site 475, Marseille
  - Boehringer Ingelheim Investigator site 476, Marseille
  - Boehringer Ingelheim Investigator site 477, Marseille
  - Boehringer Ingelheim Investigator site 478, Marseille
  - Boehringer Ingelheim Investigator site 479, Marseille
  - Boehringer Ingelheim Investigator site 480, Marseille
  - Boehringer Ingelheim Investigator site 481, Marseille
  - Boehringer Ingelheim Investigator site 482, Marseille
  - Boehringer Ingelheim Investigator site 483, Marseille
  - Boehringer Ingelheim Investigator site 484, Marseille
  - Boehringer Ingelheim Investigator site 485, Marseille
  - Boehringer Ingelheim Investigator site 486, Marseille
  - Boehringer Ingelheim Investigator site 487, Marseille
  - Boehringer Ingelheim Investigator site 488, Marseille
  - Boehringer Ingelheim Investigator site 489, Marseille
  - Boehringer Ingelheim Investigator site 490, Marseille
  - Boehringer Ingelheim Investigator site 491, Marseille
  - Boehringer Ingelheim Investigator site 492, Marseille
  - Boehringer Ingelheim Investigator site 493, Martigues
  - Boehringer Ingelheim Investigator site 494, Marvejols
  - Boehringer Ingelheim Investigator site 495, Maubourguet
  - Boehringer Ingelheim Investigator site 496, Mauguio
  - Boehringer Ingelheim Investigator site 497, Maurepas
  - Boehringer Ingelheim Investigator site 498, Mauriac
  - Boehringer Ingelheim Investigator site 499, Mayenne
  - Boehringer Ingelheim Investigator site 500, Meaux
  - Boehringer Ingelheim Investigator site 502, Mennecy
  - Boehringer Ingelheim Investigator site 503, Mensignac
  - Boehringer Ingelheim Investigator site 504, Menthon-Saint-Bernard
  - Boehringer Ingelheim Investigator site 505, Menton
  - Boehringer Ingelheim Investigator site 506, Merkwiller-Pechelbronn
  - Boehringer Ingelheim Investigator site 507, Merlevenez
  - Boehringer Ingelheim Investigator site 508, Metz
  - Boehringer Ingelheim Investigator site 509, Metz
  - Boehringer Ingelheim Investigator site 510, Metz
  - Boehringer Ingelheim Investigator site 511, Meursault
  - Boehringer Ingelheim Investigator site 512, Meyzieu
  - Boehringer Ingelheim Investigator site 513, Mezzavia
  - Boehringer Ingelheim Investigator site 501, Méjannes-lès-Alès
  - Boehringer Ingelheim Investigator site 514, Mirecourt
  - Boehringer Ingelheim Investigator site 515, Moissac
  - Boehringer Ingelheim Investigator site 516, Moncé-en-Belin
  - Boehringer Ingelheim Investigator site 517, Moncontour de Bretagne
  - Boehringer Ingelheim Investigator site 518, Monéteau
  - Boehringer Ingelheim Investigator site 519, Monéteau
  - Boehringer Ingelheim Investigator site 520, Monflanquin
  - Boehringer Ingelheim Investigator site 521, Montauban
  - Boehringer Ingelheim Investigator site 522, Montauban
  - Boehringer Ingelheim Investigator site 523, Montbéliard
  - Boehringer Ingelheim Investigator site 524, Montceau-les-Mines
  - Boehringer Ingelheim Investigator site 525, Montluçon
  - Boehringer Ingelheim Investigator site 526, Montluçon
  - Boehringer Ingelheim Investigator site 527, Montluçon
  - Boehringer Ingelheim Investigator site 528, Montluçon
  - Boehringer Ingelheim Investigator site 529, Montoire-sur-le-Loir
  - Boehringer Ingelheim Investigator site 530, Montpellier
  - Boehringer Ingelheim Investigator site 531, Montpellier
  - Boehringer Ingelheim Investigator site 532, Montpellier
  - Boehringer Ingelheim Investigator site 533, Montpellier
  - Boehringer Ingelheim Investigator site 535, Montreuil-sur-Ille
  - Boehringer Ingelheim Investigator site 536, Montrevault
  - Boehringer Ingelheim Investigator site 537, Montrevel-en-Bresse
  - Boehringer Ingelheim Investigator site 534, Montréal-la-Cluse
  - Boehringer Ingelheim Investigator site 538, Moreuil
  - Boehringer Ingelheim Investigator site 539, Morsang-sur-Orge
  - Boehringer Ingelheim Investigator site 540, Morsang-sur-Orge
  - Boehringer Ingelheim Investigator site 541, Moutiers-les-Mauxfaits
  - Boehringer Ingelheim Investigator site 542, Mulhouse
  - Boehringer Ingelheim Investigator site 544, Nancy
  - Boehringer Ingelheim Investigator site 543, Nançay
  - Boehringer Ingelheim Investigator site 545, Nangis
  - Boehringer Ingelheim Investigator site 546, Nanterre
  - Boehringer Ingelheim Investigator site 547, Nantes
  - Boehringer Ingelheim Investigator site 548, Nantes
  - Boehringer Ingelheim Investigator site 549, Nanteuil-en-Vallée
  - Boehringer Ingelheim Investigator site 550, Narbonne
  - Boehringer Ingelheim Investigator site 551, Nersac
  - Boehringer Ingelheim Investigator site 552, Neufchef
  - Boehringer Ingelheim Investigator site 553, Neuilly-lès-Dijon
  - Boehringer Ingelheim Investigator site 554, Neuilly-Plaisance
  - Boehringer Ingelheim Investigator site 555, Neuilly-sur-Seine
  - Boehringer Ingelheim Investigator site 556, Neuilly-sur-Seine
  - Boehringer Ingelheim Investigator site 557, Neuilly-sur-Seine
  - Boehringer Ingelheim Investigator site 558, Neuves-Maisons
  - Boehringer Ingelheim Investigator site 559, Neuvy-le-Roi
  - Boehringer Ingelheim Investigator site 560, Nice
  - Boehringer Ingelheim Investigator site 561, Nice
  - Boehringer Ingelheim Investigator site 562, Nice
  - Boehringer Ingelheim Investigator site 563, Nice
  - Boehringer Ingelheim Investigator site 564, Nice
  - Boehringer Ingelheim Investigator site 565, Nice
  - Boehringer Ingelheim Investigator site 566, Nice
  - Boehringer Ingelheim Investigator site 567, Nice
  - Boehringer Ingelheim Investigator site 570, Niort
  - Boehringer Ingelheim Investigator site 568, Nîmes
  - Boehringer Ingelheim Investigator site 569, Nîmes
  - Boehringer Ingelheim Investigator site 571, Noé
  - Boehringer Ingelheim Investigator site 572, Nogent-le-Rotrou
  - Boehringer Ingelheim Investigator site 573, Noisy-le-Sec
  - Boehringer Ingelheim Investigator site 574, Norrent-Fontes
  - Boehringer Ingelheim Investigator site 575, Nort-sur-Erdre
  - Boehringer Ingelheim Investigator site 576, Notre-Dame-d'Oé
  - Boehringer Ingelheim Investigator site 577, Nouan-le-Fuzelier
  - Boehringer Ingelheim Investigator site 578, Nouzonville
  - Boehringer Ingelheim Investigator site 579, Noyen-sur-Sarthe
  - Boehringer Ingelheim Investigator site 580, Noyon
  - Boehringer Ingelheim Investigator site 581, Oberhausbergen
  - Boehringer Ingelheim Investigator site 582, Obernai
  - Boehringer Ingelheim Investigator site 583, Oissel-sur-Seine
  - Boehringer Ingelheim Investigator site 584, Olby
  - Boehringer Ingelheim Investigator site 585, Ondres
  - Boehringer Ingelheim Investigator site 586, Oraison
  - Boehringer Ingelheim Investigator site 587, Orange
  - Boehringer Ingelheim Investigator site 588, Orange
  - Boehringer Ingelheim Investigator site 589, Orchamps-Vennes
  - Boehringer Ingelheim Investigator site 590, Orléans
  - Boehringer Ingelheim Investigator site 591, Orléans
  - Boehringer Ingelheim Investigator site 592, Orly
  - Boehringer Ingelheim Investigator site 593, Orry-la-Ville
  - Boehringer Ingelheim Investigator site 594, Ouistreham
  - Boehringer Ingelheim Investigator site 595, Oullins
  - Boehringer Ingelheim Investigator site 596, Oyonnax
  - Boehringer Ingelheim Investigator site 597, Paimpol
  - Boehringer Ingelheim Investigator site 598, Paimpol
  - Boehringer Ingelheim Investigator site 599, Pantin
  - Boehringer Ingelheim Investigator site 600, Paray-le-Monial
  - Boehringer Ingelheim Investigator site 601, Paray-le-Monial
  - Boehringer Ingelheim Investigator site 602, Parçay-les-Pins
  - Boehringer Ingelheim Investigator site 603, Pardies
  - Boehringer Ingelheim Investigator site 604, Parempuyre
  - Boehringer Ingelheim Investigator site 605, Parigné-l'Évêque
  - Boehringer Ingelheim Investigator site 606, Paris
  - Boehringer Ingelheim Investigator site 607, Paris
  - Boehringer Ingelheim Investigator site 608, Paris
  - Boehringer Ingelheim Investigator site 609, Paris
  - Boehringer Ingelheim Investigator site 610, Paris
  - Boehringer Ingelheim Investigator site 611, Paris
  - Boehringer Ingelheim Investigator site 612, Paris
  - Boehringer Ingelheim Investigator site 613, Paris
  - Boehringer Ingelheim Investigator site 614, Paris
  - Boehringer Ingelheim Investigator site 615, Paris
  - Boehringer Ingelheim Investigator site 616, Paris
  - Boehringer Ingelheim Investigator site 617, Paris
  - Boehringer Ingelheim Investigator site 618, Paris
  - Boehringer Ingelheim Investigator site 619, Paris
  - Boehringer Ingelheim Investigator site 620, Paris
  - Boehringer Ingelheim Investigator site 621, Paris
  - Boehringer Ingelheim Investigator site 622, Paris
  - Boehringer Ingelheim Investigator site 623, Paris
  - Boehringer Ingelheim Investigator site 624, Paris
  - Boehringer Ingelheim Investigator site 625, Paris
  - Boehringer Ingelheim Investigator site 626, Paris
  - Boehringer Ingelheim Investigator site 627, Paris
  - Boehringer Ingelheim Investigator site 628, Paris
  - Boehringer Ingelheim Investigator site 629, Paris
  - Boehringer Ingelheim Investigator site 630, Paris
  - Boehringer Ingelheim Investigator site 631, Paris
  - Boehringer Ingelheim Investigator site 632, Paris
  - Boehringer Ingelheim Investigator site 633, Paris
  - Boehringer Ingelheim Investigator site 634, Paris
  - Boehringer Ingelheim Investigator site 635, Paris
  - Boehringer Ingelheim Investigator site 636, Paris
  - Boehringer Ingelheim Investigator site 637, Paris
  - Boehringer Ingelheim Investigator site 638, Parthenay
  - Boehringer Ingelheim Investigator site 639, Pau
  - Boehringer Ingelheim Investigator site 640, Pau
  - Boehringer Ingelheim Investigator site 641, Peaugres
  - Boehringer Ingelheim Investigator site 642, Penmarch
  - Boehringer Ingelheim Investigator site 645, Perpignan
  - Boehringer Ingelheim Investigator site 646, Perpignan
  - Boehringer Ingelheim Investigator site 647, Pessac
  - Boehringer Ingelheim Investigator site 648, Peyrens
  - Boehringer Ingelheim Investigator site 649, Peyrestortes
  - Boehringer Ingelheim Investigator site 643, Péronne
  - Boehringer Ingelheim Investigator site 644, Péronne
  - Boehringer Ingelheim Investigator site 650, Pfetterhouse
  - Boehringer Ingelheim Investigator site 651, Plabennec
  - Boehringer Ingelheim Investigator site 652, Pleaux
  - Boehringer Ingelheim Investigator site 653, Pléhédel
  - Boehringer Ingelheim Investigator site 654, Plélan-le-Grand
  - Boehringer Ingelheim Investigator site 655, Ploemeur
  - Boehringer Ingelheim Investigator site 656, Plouédern
  - Boehringer Ingelheim Investigator site 657, Poitiers
  - Boehringer Ingelheim Investigator site 658, Poitiers
  - Boehringer Ingelheim Investigator site 659, Poncin
  - Boehringer Ingelheim Investigator site 660, Pont-de-Buis-lès-Quimerch
  - Boehringer Ingelheim Investigator site 661, Pontailler-sur-Saône
  - Boehringer Ingelheim Investigator site 662, Pornichet
  - Boehringer Ingelheim Investigator site 663, Port-de-Bouc
  - Boehringer Ingelheim Investigator site 664, Poussan
  - Boehringer Ingelheim Investigator site 665, Pouyastruc
  - Boehringer Ingelheim Investigator site 666, Privas
  - Boehringer Ingelheim Investigator site 667, Provins
  - Boehringer Ingelheim Investigator site 668, Provins
  - Boehringer Ingelheim Investigator site 669, Puget-Ville
  - Boehringer Ingelheim Investigator site 670, Puteaux
  - Boehringer Ingelheim Investigator site 671, Puttelange-aux-Lacs
  - Boehringer Ingelheim Investigator site 672, Puycasquier
  - Boehringer Ingelheim Investigator site 673, Quarante
  - Boehringer Ingelheim Investigator site 674, Quiberon
  - Boehringer Ingelheim Investigator site 675, Quimperlé
  - Boehringer Ingelheim Investigator site 676, Quincy-Voisins
  - Boehringer Ingelheim Investigator site 677, Rabastens-de-Bigorre
  - Boehringer Ingelheim Investigator site 678, Rambouillet
  - Boehringer Ingelheim Investigator site 679, Rebais
  - Boehringer Ingelheim Investigator site 680, Rennes
  - Boehringer Ingelheim Investigator site 681, Rennes
  - Boehringer Ingelheim Investigator site 682, Rezé
  - Boehringer Ingelheim Investigator site 683, Riedisheim
  - Boehringer Ingelheim Investigator site 684, Rieupeyroux
  - Boehringer Ingelheim Investigator site 685, Rigney
  - Boehringer Ingelheim Investigator site 686, Rilhac-Rancon
  - Boehringer Ingelheim Investigator site 687, Rodez
  - Boehringer Ingelheim Investigator site 688, Rodez
  - Boehringer Ingelheim Investigator site 689, Rodez
  - Boehringer Ingelheim Investigator site 690, Rognes
  - Boehringer Ingelheim Investigator site 691, Roissy-en-France
  - Boehringer Ingelheim Investigator site 692, Rombas
  - Boehringer Ingelheim Investigator site 693, Romorantin-Lanthenay
  - Boehringer Ingelheim Investigator site 694, Ronchamp
  - Boehringer Ingelheim Investigator site 695, Roncq
  - Boehringer Ingelheim Investigator site 696, Roncq
  - Boehringer Ingelheim Investigator site 697, Roquevaire
  - Boehringer Ingelheim Investigator site 698, Rosières-en-Santerre
  - Boehringer Ingelheim Investigator site 699, Rosny-sous-Bois
  - Boehringer Ingelheim Investigator site 700, Roubaix
  - Boehringer Ingelheim Investigator site 701, Rouillac
  - Boehringer Ingelheim Investigator site 702, Roulans
  - Boehringer Ingelheim Investigator site 703, Ruoms
  - Boehringer Ingelheim Investigator site 704, Sainpuits
  - Boehringer Ingelheim Investigator site 705, Sains-du-Nord
  - Boehringer Ingelheim Investigator site 706, Sains-du-Nord
  - Boehringer Ingelheim Investigator site 782, Saint Maximin La Ste Baume
  - Boehringer Ingelheim Investigator site 798, Saint Rene Hillion
  - Boehringer Ingelheim Investigator site 737, Saint-Aigulin
  - Boehringer Ingelheim Investigator site 738, Saint-Amand-Montrond
  - Boehringer Ingelheim Investigator site 739, Saint-André-les-Vergers
  - Boehringer Ingelheim Investigator site 740, Saint-André-lez-Lille
  - Boehringer Ingelheim Investigator site 741, Saint-Aubin-des-Châteaux
  - Boehringer Ingelheim Investigator site 742, Saint-Avertin
  - Boehringer Ingelheim Investigator site 743, Saint-Avold
  - Boehringer Ingelheim Investigator site 744, Saint-Avold
  - Boehringer Ingelheim Investigator site 745, Saint-Avold
  - Boehringer Ingelheim Investigator site 746, Saint-Avold
  - Boehringer Ingelheim Investigator site 747, Saint-Barthélémy
  - Boehringer Ingelheim Investigator site 748, Saint-Benoît
  - Boehringer Ingelheim Investigator site 749, Saint-Brieuc
  - Boehringer Ingelheim Investigator site 750, Saint-Chamond
  - Boehringer Ingelheim Investigator site 751, Saint-Chamond
  - Boehringer Ingelheim Investigator site 752, Saint-Clément
  - Boehringer Ingelheim Investigator site 753, Saint-Cyr-sur-Mer
  - Boehringer Ingelheim Investigator site 754, Saint-Didier-en-Velay
  - Boehringer Ingelheim Investigator site 755, Saint-Dié
  - Boehringer Ingelheim Investigator site 756, Saint-Dié
  - Boehringer Ingelheim Investigator site 757, Saint-Dizier
  - Boehringer Ingelheim Investigator site 758, Saint-Dizier
  - Boehringer Ingelheim Investigator site 759, Saint-Estève
  - Boehringer Ingelheim Investigator site 760, Saint-Etienne
  - Boehringer Ingelheim Investigator site 761, Saint-Etienne
  - Boehringer Ingelheim Investigator site 762, Saint-Étienne-de-Montluc
  - Boehringer Ingelheim Investigator site 763, Saint-Étienne-du-Rouvray
  - Boehringer Ingelheim Investigator site 764, Saint-Georges-de-Didonne
  - Boehringer Ingelheim Investigator site 765, Saint-Germain-de-la-Coudre
  - Boehringer Ingelheim Investigator site 766, Saint-Guénolé
  - Boehringer Ingelheim Investigator site 767, Saint-Hilaire-lez-Cambrai
  - Boehringer Ingelheim Investigator site 768, Saint-Jean-de-Luz
  - Boehringer Ingelheim Investigator site 769, Saint-Jean-le-Blanc
  - Boehringer Ingelheim Investigator site 770, Saint-Julien-de-Concelles
  - Boehringer Ingelheim Investigator site 771, Saint-Julien-les-Rosiers
  - Boehringer Ingelheim Investigator site 772, Saint-Laurent-du-Var
  - Boehringer Ingelheim Investigator site 773, Saint-Laurent-du-Var
  - Boehringer Ingelheim Investigator site 774, Saint-Laurent-sur-Sèvre
  - Boehringer Ingelheim Investigator site 775, Saint-Loup-sur-Semouse
  - Boehringer Ingelheim Investigator site 776, Saint-Lyé
  - Boehringer Ingelheim Investigator site 777, Saint-Lyé
  - Boehringer Ingelheim Investigator site 779, Saint-Marcellin
  - Boehringer Ingelheim Investigator site 780, Saint-Martin-de-Seignanx
  - Boehringer Ingelheim Investigator site 781, Saint-Martin-le-Beau
  - Boehringer Ingelheim Investigator site 783, Saint-Médard-en-Jalles
  - Boehringer Ingelheim Investigator site 784, Saint-Médard-en-Jalles
  - Boehringer Ingelheim Investigator site 785, Saint-Nazaire
  - Boehringer Ingelheim Investigator site 787, Saint-Nicolas en Forêt
  - Boehringer Ingelheim Investigator site 786, Saint-Nicolas-de-Port
  - Boehringer Ingelheim Investigator site 788, Saint-Omer
  - Boehringer Ingelheim Investigator site 789, Saint-Orens-de-Gameville
  - Boehringer Ingelheim Investigator site 790, Saint-Ouen
  - Boehringer Ingelheim Investigator site 791, Saint-Pierre-en-Val
  - Boehringer Ingelheim Investigator site 792, Saint-Pol-de-Léon
  - Boehringer Ingelheim Investigator site 793, Saint-Pol-sur-Mer
  - Boehringer Ingelheim Investigator site 794, Saint-Priest
  - Boehringer Ingelheim Investigator site 795, Saint-Quentin
  - Boehringer Ingelheim Investigator site 796, Saint-Rambert-d'Albon
  - Boehringer Ingelheim Investigator site 797, Saint-Rémy-lès-Chevreuse
  - Boehringer Ingelheim Investigator site 799, Saint-Saëns
  - Boehringer Ingelheim Investigator site 800, Saint-Saëns
  - Boehringer Ingelheim Investigator site 801, Saint-Sauveur
  - Boehringer Ingelheim Investigator site 802, Saint-Sébastien-sur-Loire
  - Boehringer Ingelheim Investigator site 803, Saint-Vrain
  - Boehringer Ingelheim Investigator site 707, Saints
  - Boehringer Ingelheim Investigator site 708, Salbris
  - Boehringer Ingelheim Investigator site 709, Salles
  - Boehringer Ingelheim Investigator site 710, Salomé
  - Boehringer Ingelheim Investigator site 711, Samer
  - Boehringer Ingelheim Investigator site 712, Sarcelles
  - Boehringer Ingelheim Investigator site 713, Sarlat-la-Canéda
  - Boehringer Ingelheim Investigator site 714, Sarras
  - Boehringer Ingelheim Investigator site 715, Sarrebourg
  - Boehringer Ingelheim Investigator site 716, Sarreguemines
  - Boehringer Ingelheim Investigator site 717, Sarreguemines
  - Boehringer Ingelheim Investigator site 718, Savigny-sur-Orge
  - Boehringer Ingelheim Investigator site 719, Savigny-sur-Orge
  - Boehringer Ingelheim Investigator site 720, Savigny-sur-Orge
  - Boehringer Ingelheim Investigator site 721, Schiltigheim
  - Boehringer Ingelheim Investigator site 722, Sedan
  - Boehringer Ingelheim Investigator site 724, Seraincourt
  - Boehringer Ingelheim Investigator site 727, Sers
  - Boehringer Ingelheim Investigator site 730, Sevran
  - Boehringer Ingelheim Investigator site 731, Seysses
  - Boehringer Ingelheim Investigator site 728, Sète
  - Boehringer Ingelheim Investigator site 729, Sète
  - Boehringer Ingelheim Investigator site 723, Sélestat
  - Boehringer Ingelheim Investigator site 725, Sérignan
  - Boehringer Ingelheim Investigator site 726, Sérignan
  - Boehringer Ingelheim Investigator site 732, Sisteron
  - Boehringer Ingelheim Investigator site 733, Six-Fours-les-Plages
  - Boehringer Ingelheim Investigator site 734, Six-Fours-les-Plages
  - Boehringer Ingelheim Investigator site 735, Soisy-sous-Montmorency
  - Boehringer Ingelheim Investigator site 736, Soyaux
  - Boehringer Ingelheim Investigator site 778, St-Malo
  - Boehringer Ingelheim Investigator site 804, Stains
  - Boehringer Ingelheim Investigator site 805, Ste Cecile
  - Boehringer Ingelheim Investigator site 806, Ste Fereole
  - Boehringer Ingelheim Investigator site 807, Ste Hermine
  - Boehringer Ingelheim Investigator site 808, Ste Mere Eglise
  - Boehringer Ingelheim Investigator site 809, Ste Savine
  - Boehringer Ingelheim Investigator site 810, Strasbourg
  - Boehringer Ingelheim Investigator site 811, Strasbourg
  - Boehringer Ingelheim Investigator site 812, Strasbourg
  - Boehringer Ingelheim Investigator site 813, Sucy-en-Brie
  - Boehringer Ingelheim Investigator site 814, Suresnes
  - Boehringer Ingelheim Investigator site 815, Tarascon
  - Boehringer Ingelheim Investigator site 816, Tarascon-sur-Ariège
  - Boehringer Ingelheim Investigator site 817, Tarbes
  - Boehringer Ingelheim Investigator site 818, Tarnos
  - Boehringer Ingelheim Investigator site 819, Taverny
  - Boehringer Ingelheim Investigator site 820, Ternay
  - Boehringer Ingelheim Investigator site 821, Terrasson La Villedieu
  - Boehringer Ingelheim Investigator site 822, Tessy-sur-Vire
  - Boehringer Ingelheim Investigator site 823, Teyran
  - Boehringer Ingelheim Investigator site 824, Thaon
  - Boehringer Ingelheim Investigator site 825, Thionville
  - Boehringer Ingelheim Investigator site 826, Thouaré-sur-Loire
  - Boehringer Ingelheim Investigator site 827, Tilly-sur-Seulles
  - Boehringer Ingelheim Investigator site 828, Torcy
  - Boehringer Ingelheim Investigator site 829, Toufflers
  - Boehringer Ingelheim Investigator site 830, Toulon
  - Boehringer Ingelheim Investigator site 831, Toulon
  - Boehringer Ingelheim Investigator site 832, Toulon
  - Boehringer Ingelheim Investigator site 833, Toulouse
  - Boehringer Ingelheim Investigator site 834, Toulouse
  - Boehringer Ingelheim Investigator site 835, Toulouse
  - Boehringer Ingelheim Investigator site 836, Tourcoing
  - Boehringer Ingelheim Investigator site 837, Tourcoing
  - Boehringer Ingelheim Investigator site 838, Tournon-sur-Rhône
  - Boehringer Ingelheim Investigator site 839, Tours
  - Boehringer Ingelheim Investigator site 841, Trets
  - Boehringer Ingelheim Investigator site 840, Trélazé
  - Boehringer Ingelheim Investigator site 842, Trévières
  - Boehringer Ingelheim Investigator site 843, Triel-sur-Seine
  - Boehringer Ingelheim Investigator site 844, Troissereux
  - Boehringer Ingelheim Investigator site 845, Troyes
  - Boehringer Ingelheim Investigator site 846, Unieux
  - Boehringer Ingelheim Investigator site 847, Ussac
  - Boehringer Ingelheim Investigator site 848, Vailly-sur-Aisne
  - Boehringer Ingelheim Investigator site 849, Valenton
  - Boehringer Ingelheim Investigator site 850, Vallauris
  - Boehringer Ingelheim Investigator site 851, Valras-Plage
  - Boehringer Ingelheim Investigator site 852, Valréas
  - Boehringer Ingelheim Investigator site 853, Vanves
  - Boehringer Ingelheim Investigator site 854, Vars
  - Boehringer Ingelheim Investigator site 856, Venarey-les-Laumes
  - Boehringer Ingelheim Investigator site 858, Vendôme
  - Boehringer Ingelheim Investigator site 859, Vendôme
  - Boehringer Ingelheim Investigator site 857, Vendœuvres
  - Boehringer Ingelheim Investigator site 860, Verdun
  - Boehringer Ingelheim Investigator site 862, Verfeil
  - Boehringer Ingelheim Investigator site 863, Vern-sur-Seiche
  - Boehringer Ingelheim Investigator site 864, Verrières-le-Buisson
  - Boehringer Ingelheim Investigator site 865, Versailles
  - Boehringer Ingelheim Investigator site 866, Vert-Saint-Denis
  - Boehringer Ingelheim Investigator site 867, Vesoul
  - Boehringer Ingelheim Investigator site 855, Vélizy-Villacoublay
  - Boehringer Ingelheim Investigator site 861, Véretz
  - Boehringer Ingelheim Investigator site 868, Vézénobres
  - Boehringer Ingelheim Investigator site 869, Vias
  - Boehringer Ingelheim Investigator site 870, Vichy
  - Boehringer Ingelheim Investigator site 871, Vichy
  - Boehringer Ingelheim Investigator site 872, Vichy
  - Boehringer Ingelheim Investigator site 873, Vif
  - Boehringer Ingelheim Investigator site 874, Vihiers
  - Boehringer Ingelheim Investigator site 875, Ville-di-Pietrabugno
  - Boehringer Ingelheim Investigator site 876, Villeblevin
  - Boehringer Ingelheim Investigator site 877, Villefranche-de-Rouergue
  - Boehringer Ingelheim Investigator site 878, Villefranche-de-Rouergue
  - Boehringer Ingelheim Investigator site 879, Villefranche-sur-Saône
  - Boehringer Ingelheim Investigator site 880, Villefranche-sur-Saône
  - Boehringer Ingelheim Investigator site 881, Villejuif
  - Boehringer Ingelheim Investigator site 882, Villemeux-sur-Eure
  - Boehringer Ingelheim Investigator site 883, Villenave-d'Ornon
  - Boehringer Ingelheim Investigator site 884, Villeneuve-sur-Lot
  - Boehringer Ingelheim Investigator site 885, Villeneuve-sur-Lot
  - Boehringer Ingelheim Investigator site 886, Villepreux
  - Boehringer Ingelheim Investigator site 887, Villepreux
  - Boehringer Ingelheim Investigator site 888, Villers-lès-Nancy
  - Boehringer Ingelheim Investigator site 889, Villerupt
  - Boehringer Ingelheim Investigator site 890, Villette-de-Vienne
  - Boehringer Ingelheim Investigator site 891, Villeurbanne
  - Boehringer Ingelheim Investigator site 892, Villeurbanne
  - Boehringer Ingelheim Investigator site 893, Villeurbanne
  - Boehringer Ingelheim Investigator site 894, Villeurbanne
  - Boehringer Ingelheim Investigator site 895, Villeurbanne
  - Boehringer Ingelheim Investigator site 896, Villiers-le-Bel
  - Boehringer Ingelheim Investigator site 897, Villiers-sur-Orge
  - Boehringer Ingelheim Investigator site 898, Vitrolles
  - Boehringer Ingelheim Investigator site 899, Vitrolles
  - Boehringer Ingelheim Investigator site 900, Vitry-sur-Seine
  - Boehringer Ingelheim Investigator site 901, Vivier-au-Court
  - Boehringer Ingelheim Investigator site 902, Viviers
  - Boehringer Ingelheim Investigator site 903, Vrigne-aux-Bois
  - Boehringer Ingelheim Investigator site 904, Wallers
  - Boehringer Ingelheim Investigator site 905, Wambrechies
  - Boehringer Ingelheim Investigator site 906, Wambrechies
  - Boehringer Ingelheim Investigator site 907, Wattignies
  - Boehringer Ingelheim Investigator site 908, Wattignies
  - Boehringer Ingelheim Investigator site 909, Wattrelos
  - Boehringer Ingelheim Investigator site 910, Wattrelos
  - Boehringer Ingelheim Investigator site 911, Weitbruch
  - Boehringer Ingelheim Investigator site 912, Wingles
  - Boehringer Ingelheim Investigator site 913, Wittisheim
  - Boehringer Ingelheim Investigator site 914, Ydes
  - Boehringer Ingelheim Investigator site 915, Zillisheim

RESULTS

PARTICIPANT FLOW:
Groups:
- Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg: Patients treated at least 8 weeks with Fixed Dose Combination (FDC)
Period: Overall Study
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Started | 2411
Completed | 1994
Not Completed | 417
Not completed — Protocol Violation | 187
Not completed — Non-evaluable Subjects | 230

BASELINE CHARACTERISTICS:
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 1994
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 835
  Male | 1159
Hypertension treatments prescribed prior to initiation of treatment [Number; unit: Percentage of participants] — Hypertension treatments prescribed prior to initiation of treatment with telmisartan 80mg in a FDC with HCTZ 25 mg
  Percentage of participants
    Angiotensin II antagonist | 71.8
    Diuretic | 64.3
    Calcium channel blocker | 23.3
    Beta-blocker | 20.5
Conditions for prescribing 80 mg telmisartan in fixed combination with 25 mg HCTZ [Number; unit: Percentage of participants] — Conditions for prescribing 80 mg telmisartan in fixed combination with 25 mg HCTZ were ,
  "Lack of efficacy of previous treatments" and "To decrease the number of treatment administration throughout the day"
  Percentage of participants
    Lack of efficacy | 53.8
    To decrease the number of treatment | 33.1
Cardiovascular risk factors (including the existence of a metabolic syndrome) [Number; unit: Percentage of participants] — Number of Patients used in the analysis for Cardiovascular risk factors (including the existence of a metabolic syndrome) were 322 Participants with existence of a metabolic syndrome
  Percentage of participants
    Age (male>50 or female>60) | 82.0
    Smoking | 23.9
    Family History | 28.9
    Diabetes | 54.3
    LDL-Cholesterol ≥ 1.6 g/L | 72.4
    HDL-Cholesterol ≤ 0.4 g/L | 20.5

OUTCOME MEASURES:

1. Primary Outcome: Rate of BP Control in Hypertensive Patients
Description: Percentage of controlled Patients at the Study End.
  Control rate of hypertension in general practice and in cardiology defined as systolic blood pressure (SBP) and diastolic blood pressure (DBP) <140/90 mmHg for unselected hypertensive patients and SBP and DBP <130/80 mmHg for hypertensive patients at high cardiovascular risk (patients with diabetes and patients with impaired renal function) as defined in the recommendations of the French National Health Authority (HAS) 2005 guidelines.
Time Frame: Baseline to a minimum of 8 weeks of treatment
Population: Descriptive statistical analysis was performed for the entire study population on the FAS in intention-to-treat (ITT) as well as on the Per protocol set (PPS) in per protocol (PP). The difference between the numbers of patients was inferior than 10% ; the results of the primary objective was presented in PPS.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 1994
Percentage of Participants | 51.3 [49.0 to 53.5]

2. Secondary Outcome: Systolic Blood Pressure (SBP) After at Least 8 Weeks of Treatment in Overall Study Population
Description: Mean SBP measured at the Study End
Time Frame: baseline to a minimum of 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 1994
mm Hg | 137.3 (9.6)

3. Secondary Outcome: Diastolic Blood Pressure (DBP) After at Least 8 Weeks of Treatment in Overall Study Population
Description: Mean DBP measured at the Study End
Time Frame: baseline to a minimum of 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 1994
mm Hg | 80.1 (7.2)

4. Secondary Outcome: Systolic Blood Pressure (SBP) After at Least 8 Weeks of Treatment in Population at High Cardiovascular Risk
Description: Mean SBP measured at the Study End
Time Frame: baseline to a minimum of 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 972
mmHg | 144.3 (7.9)

5. Secondary Outcome: Diastolic Blood Pressure (DBP) After at Least 8 Weeks of Treatment in Population at High Cardiovascular Risk
Description: Mean DBP measured at the Study End
Time Frame: baseline to a minimum of 8 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 972
mmHg | 82.9 (7.2)

6. Secondary Outcome: Rate of BP Control by Risk Factor According to the Recommendations ESH/ESC 2007
Description: The proportion of patients with blood pressure (BP) control, per risk factor. High risk factors determined according to the recommendations of the ESH/ESC 2007.
Time Frame: Baseline to a minimum of 8 weeks of treatment
Population: Per protocol set (PPS)
Measure: Number; unit: percentage of patients
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Number analyzed (Participants) | 661
percentage of patients
  Age >60 years | 51.9 [99.4 to 100]
  Diabetes | 5.0 [18.3 to 24.7]
  Renal Failure | 3.8
  History of TIA/CVA | 3.9
  Coronary Chronic Disease | 8.3

ADVERSE EVENTS:
Time Frame: 6 months
Description: Study duration between first included and last included patients.
Arm/Group | Telmisartan (T) 80mg/Hydrochlorothiazide (HCTZ) 25 mg
Serious Adverse Events (participants affected / at risk) | 0/1994
Other Adverse Events (participants affected / at risk) | 0/1994

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.